CLINICAL TRIAL: NCT03562455
Title: Assessing the Effectiveness of Virtual Reality for Power Wheelchair Driving Training
Brief Title: Virtual Reality for Power Wheelchair Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Brad Dicianno, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRO18010297
Record Dates: First submitted 2018-05-22; First posted 2018-06-19 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Spinal Diseases
Keywords: Virtual Reality; Wheelchairs
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Intervention Model Description: The study will contain two arms. One group will receive virtual reality power wheelchair training, and the other will receive in-person wheelchair training by a therapist.
Who Masked: Outcomes Assessor
Masking Description: The individual assessing performance outcomes will not be aware of which intervention the participants received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Training (Experimental): Participants will receive virtual reality power wheelchair training using VRSim 3.0 in this group.
  Interventions: Other: VRSim 3.0
- In-person Therapist Training (Active Comparator): Participants will receive in-person wheelchair training by a therapist in this group.
  Interventions: Behavioral: In-Person Wheelchair Training

INTERVENTIONS:
Other: VRSim 3.0 — VRSim 3.0 is a virtual reality training module.
  Arms: Virtual Reality Training
Behavioral: In-Person Wheelchair Training — A therapist will be used to train power wheelchair users.
  Arms: In-person Therapist Training

SUMMARY:
The objective of this study is to evaluate the impact of VRSim 3.0 on power wheelchair (PWC) driving skills and to obtain qualitative feedback from users on the design of the virtual reality (VR) simulator to inform device development.

DETAILED DESCRIPTION:
A virtual reality platform may lead to better training of people with complex disabilities who desire to be power wheelchair users and thus allow them to benefit from living a more active life. A virtual reality training program could significantly impact the lives of people with disabilities by improving function, reducing abandonment of power wheelchairs, and reducing morbidity and mortality and associated costs occurring from power wheelchair accidents. This new virtual reality training program will reflect improvements in accessibility, customization, simulator sickness, ease of use, and will have report generating capabilities as compared to previous virtual reality training platforms. The investigators expect that virtual reality training will be a superior alternative to standard in-person wheelchair training.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must be 14 years or older.
* Volunteers must have a disability that prevents them from effectively and independently using a manual wheelchair, power assist wheelchair, or scooter.
* Volunteers must be able to communicate in English, follow simple commands, and give written informed consent.

Exclusion Criteria:

* Volunteers with active seizures.
* Volunteers who have active pelvic or thigh wounds.
* Volunteers who require a test wheelchair but who exceed the weight capacity of the test wheelchair (>300 lbs).
* Volunteers who require a test wheelchair but also require specialized seating that cannot be replicated for the training.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Power Wheelchair Driving Skill | This outcome measure will be assessed at each of 4 training sessions, which may take up to one year to complete.
  Power wheelchair driving skills will be evaluated using the Power Mobility Clinical Driving Assessment (PMCDA). The PMCDA contains 23 questions related to specific power wheelchair driving tasks. Each task will be given a score from 1 to 3; a score of 1 will be given if the driver requires physical assistance or cannot complete the task, a score of 2 will be given if the driver requires verbal or auditory hints or cues, but no physical assistance, and a score of 3 will be given if the driver completes the task without help. Scores will be added together for a possible total from 23 to 69.

SECONDARY OUTCOMES:
Perception of Virtual Reality Training System | This outcome measure will be assessed at the completion of the study, which may take up to one year to complete.
  Qualitative feedback on the participants' experience with VRSim 3.0 will be obtained to inform future software development using a semi-structured interview as well as a Virtual Experience Test (VET) survey. The semi-structured interview will contain open-ended questions aimed at exploring usability factors that may be barriers or facilitators to the use of VR for PWC driving training. The VET is a validated survey instrument that will be used to measure the virtual environment experience. It will contain 17 questions based on based upon five dimensions of experiential design: sensory, cognitive, affective, active, and relational. The survey questions will be scored from 1 (strongly disagree) to 5 (strongly agree).
Simulator Sickness | This outcome measure will be assessed at the beginning and end of 4 training sessions, which may take up to one year to complete.
  Participants in the virtual reality group will be given a Simulator Sickness Questionnaire (SSQ) at the beginning and end of each training session to assess the degree of simulator sickness induced by the gaming platform. The SSQ contains 16 questions based on symptoms of simulator sickness, and participants will rate each symptom as either none, slight, moderate, or severe.
Perceived Workload of Training | This outcome measure will be assessed at each of 4 training sessions, which may take up to one year to complete.
  Participants will be given a NASA-Task Load Index (NASA-TLX) survey to assess perceived workload at the end of each training session. The NASA-TLX contains 6 questions to assess workload on a scale from low to high.
Power Wheelchair Driving Capacity | This outcome measure will be measured at the beginning and end of the study, which may take up to one year to complete.
  Participants will be evaluated using the Power Mobility Screening Tool (PMST) to assess driving capacity. The PMST contains 5 questions based on motor, sensory, and cognitive skills. The questions will be scored from 1 to 3, and will be added together for a possible total from 5 to 15.

CONTACTS AND LOCATIONS:
Overall Officials: Brad E Dicianno, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Human Engineering Research Laboratories, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No